CLINICAL TRIAL: NCT07212296
Title: Robotic-Assisted Versus Conventional Total Knee Arthroplasty: A Randomized Controlled Trial With 2-Year Follow-Up
Brief Title: Randomized Controlled Trial Comparing Robotic-Assisted Versus Conventional Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Terrassa (Other)
Responsible Party: Principal Investigator, Javier Alonso, Knee Unit Surgeon, Hospital de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-21-105-058
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Knee Arthroplasty, Total; Robotic Assisted Arthroplasty; Arthropathy of Knee
Keywords: Robotic; Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional total knee replacement (Placebo Comparator): PAtietns undergoing conventional TKR
  Interventions: Procedure: Conventional total knee replacement
- Robotic TKR (Experimental): PAtietns undergoing robotic TKR
  Interventions: Procedure: Robotic TKR

INTERVENTIONS:
Procedure: Conventional total knee replacement — Knee replacement without robotic technology
  Arms: Conventional total knee replacement
Procedure: Robotic TKR — Total knee replacement WITH robotic technology
  Arms: Robotic TKR

SUMMARY:
To evaluate whether patients undergoing robotic-assisted TKA achieve better clinical-functional, radiological, and satisfaction outcomes compared with those undergoing the conventional technique, and whether operative time and complications do not increase significantly

DETAILED DESCRIPTION:
To compare clinical, functional, quality-of-life, and radiological outcomes between robotic-assisted total knee arthroplasty (RA-TKA) and conventional total knee arthroplasty (C-TKA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee arthropaty recquiring TKR

Exclusion Criteria:

* Cognitive disease
* Deformity greater than 15º of varus or 10º of valgus
* Postraumatic arthritis
* Inflamatory disease
* Other than "Persona PS" implant design
* Previus surgery

Ages: 54 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
IKDC | 2 years follow up after surgery
  standardized international system for documenting and evaluating knee problems. The IKDC Subjective Knee Form is a patient-reported outcome measure that was developed to assess both surgical and non-surgical outcomes across a wide range of knee conditions and treatment approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Alonso-Rodriguez Piedra, Orthopaedic Surgeon, MdPhD, Principal Investigator — Hospital de Terrassa
Locations (1):
- Hospital de Terrassa - Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No